CLINICAL TRIAL: NCT02150421
Title: Impact of School Curriculum Engaging Electronic Devices on Myopia Development and Progression in Primary Schoolchildren
Brief Title: Impact of Electronic Devices on Myopia Development and Progression
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Carly Lam, Professor, The Hong Kong Polytechnic University
Other Study IDs: TWGHs; TWGHs2013 (Other Grant/Funding Number: Tung Wah Group of Hospitals)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- e-book: study the course materials by using e-book

SUMMARY:
The aim of the stuy is to investigate the effects of the adoption of a curriculum with electronic devices for teaching materials and textbooks in Hong Kong schoolchildren on their changes in refractive error and visual function.

DETAILED DESCRIPTION:
With the blooming of information technology and electronic engineering in recent years, e-books or tablet computers have been introduced at some local primary and secondary schools and have been provided for their students during studying at school and at home. Parents and teachers' utmost concern are adverse effects on eye-sight of children, especially the higher progression rate in myopia and the visual discomfort which may be caused by the e-book technology.

This is a prospective cohort study to determine if implementation of electronic devices for teaching promotes myopia development and progression and affects visual function in primary schoolchildren.

The schools will introduce e-books to their students in some classes. Signed informed consent letters from parents will be obtained prior to subject recruitment and data collection. Eye examination and data collection will be conducted in primary school campus. The children from two local primary schools in same grade will be assigned into two groups by their schools. One group will use e-books (e-book group) to study course materials assigned by their teachers whereas another group will use ordinary textbooks (control group). Their refractive errors, axial length (AXL) and binocular functions will be measured and monitored at six-month intervals for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* study local primary schools

Exclusion Criteria:

* with any ocular diseases and binocular anomalies might affect visual functions or refractive development
* with history of eye surgery
* have undertaken any kind of myopia control treatment, such as bifocal lenses, orth-K, eyedrops (e.g. atropine)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary schoolchildren in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in refractive errors | 2 years
  cycloplegic autorefraction

SECONDARY OUTCOMES:
changes in axial length | 2 years
  measured by the Zeiss IOLMaster after cycloplegia
Keratometric changes | 2 years

OTHER OUTCOMES:
Phoria at distance and near | every 6-month
  Howell phoria cards

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, Professor, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No